CLINICAL TRIAL: NCT05251935
Title: Effects of Foot Muscle Exercise on Gross Motor Function and Balance Among Pes Planus Down Syndrome Patients
Brief Title: Down Syndrome and Effects of Foot Muscle Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Nazia Adeeb, Head of Department, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nazia Adeeb
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pes Planus Down Syndrome Patients
Keywords: Down syndrome; foot deformities; muscle hypotonia; pes planus; joint laxity; exercise training
MeSH Terms: conditions — Down Syndrome; Foot Deformities; Muscle Hypotonia; Flatfoot; Joint Instability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Muscle Exercise (Experimental)
  Interventions: Other: Foot Muscle Exercise Protocol
- Arch Support Insole and One Leg Balance Activities (Active Comparator)
  Interventions: Combination Product: Arch Support Insole and One Leg Balance Activities

INTERVENTIONS:
Other: Foot Muscle Exercise Protocol — Foot Muscle Exercise was given for 3 days per week for 40 minutes for the period of 6 months including home program
  Arms: Foot Muscle Exercise
Combination Product: Arch Support Insole and One Leg Balance Activities — Arch Support Insoles were provided that the child had to wear for 5 hours per day thrice weekly for 6 months plus performed one leg balance activities
  Arms: Arch Support Insole and One Leg Balance Activities

SUMMARY:
Down syndrome (DS) is a common chromosomal pediatric disorder and accounts for approximately 8 % of all congenital anomalies. Children with DS experience delays in Cognitive, Physical, Speech and Language development. Hypotonity and laxity that is part of its features causes delay on motor acquisition. Furthermore it causes musculoskeletal issues and lower extremity malalignment resulting in inefficient and abnormal pattern of movement compromising locomotion and day to day functions therefore, problems for the population further aggravates. Combined effects of these factors causes a high level of stress on foot as it provides the foundation for whole body therefore, individuals with Down syndrome are at risk for foot alignment problems. Pes planus being the most common amongst them and accounts for 91% of the total DS patients diagnosed. Pes planus causes alteration in foot kinetics and kinematics that not only interferes significantly with normal daily life activities as balance and gait but also increases the risk of musculoskeletal injuries. Hence researchers have shown interest in addressing this condition for the effective management of DS population. Conventional treatment approach are the use of insoles, foot orthosis and arch taping however, they fail to produce residual effect. Hence the present study is to determine the role of foot muscles exercises in Down Syndrome having pes planus since its effects are positively recorded in normal population.

ELIGIBILITY:
Inclusion Criteria:

* • Clinically diagnosed cases of DS including both male and female.

  * Bilateral flexible pes planus on the basis of Navicular Drop Test.
  * Able to follow instructions and adhere to the exercise program.
  * Ambulating independently.

Exclusion Criteria:

* • Visual or auditory impairment.

  * Lower limb trauma or surgical intervention past six months.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function | Baseline
  Gross Motor Function was assessed using GMFM-88 Dimensions D and E
Gross Motor Function | 12 weeks
  Gross Motor Function was assessed using GMFM-88 Dimensions D and E
Gross Motor Function | 24 weeks
  Gross Motor Function was assessed using GMFM-88 Dimensions D and E
Balance | Baseline
  Balance was assessed using Pediatric Balance Scale
Balance | 12 weeks
  Balance was assessed using Pediatric Balance Scale
Balance | 24 weeks
  Balance was assessed using Pediatric Balance Scale

CONTACTS AND LOCATIONS:
Locations (1):
- ACELP (Institute of Child Development), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No